CLINICAL TRIAL: NCT01978756
Title: Outpatient Clinic to Evaluate Late Outcome in Patients Curatively Treated for Breast Carcinoma in MAASTRO Clinic.
Brief Title: Outpatient Clinic for Late Outcome for Breast Carcinoma in MAASTRO Clinic.
Status: Completed | Type: Observational
Sponsor: Maastricht Radiation Oncology (Other)
Responsible Party: Sponsor
Other Study IDs: 12-25-15/08
Record Dates: First submitted 2013-09-02; First posted 2013-11-07 (Estimated); Last update posted 2016-05-24 (Estimated); Status verified 2016-05

CONDITIONS: Breast Cancer
Keywords: Outpatient clinic; Breast cancer; Late toxicity
MeSH Terms: conditions — Breast Neoplasms | interventions — Ambulatory Care Facilities

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — As part of the study a blood sample or saliva will be obtained, if the patient has given written informed consent to participate in the Biobank. The purpose to determine, by means of DNA and protein analysis, the relationship between DNA and protein profiles and a number of endpoints, which are important for the patient such as overall survival and side effects.
  For detailed information: ClinicalTrials.gov Identifier: NCT01084785
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Outpatient clinic: All patients treated for breast cancer with curative intent in MAASTRO clinic in 2002-2003 who are still alive, who respond to our invitation letter and are willing to participate to visit the outpatient clinic. These patients will be sent a questionnaire with both basic and more detailed questions on their disease-status and on quality of life related outcome. In addition they will be asked to come to MAASTRO clinic for a more detailed evaluation of late side effects of the treatment. Patients are seen by a physician or a physician assistant at the outpatient clinic.
  Interventions: Other: Outpatient clinic

INTERVENTIONS:
Other: Outpatient clinic — The participants are seen at the outpatient clinic by a physician or a physician assistant. To analyse fibrosis clinical examination of the breast will be performed. To analyse shoulder function anteversion / retroversion, abduction / adduction and internal / external rotation will be measured. To analyse edema the arm circumference will be measured 15 cm above and below the medial epicondyle (both sides). Also, a photograph of the breast will be made for cosmetic analysis using standardized procedures. Finally a blood sample or saliva will be obtained, if the patient has given written informed consent to participate in the Biobank.

SUMMARY:
In order to evaluate the late outcome in patients curatively treated for breast cancer, a special outpatient clinic will be developed.

There are two main purposes of the outpatient clinic. The first purpose is evaluating the results of the radiation treatment by mapping A) late toxicity and B) tumour control and survival.

The second purpose is that this outpatient clinic for late outcome will also function as a pilot for a new CAT (Computer Assisted Theragnostics, abbreviated CAT project) in which multiple late outcome variables will be recorded. In this pilot we want to investigate whether physical presence of the patient on the outpatient clinic, allowing physical examination, has any added value to the questionnaires filled in by the patient at home.

The ultimate aim of this new CAT project is to use these multicentric data to develop models for predicting both oncological outcome and late side effects. Insight in the beneficial and adverse effects of a certain treatment using these predictive models, will be required choose the optimal treatment for the individual patient using a shared decision making process.

ELIGIBILITY:
Inclusion Criteria:

* All patients treated for breast cancer with curative intent in MAASTRO clinic in 2002-2003 who are still alive.
* Consent to invitation letter and willing to participate.

Exclusion Criteria:

* Treatment without curative intent.
* No consent to invitation letter

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants are all patients who have been treated for breast cancer with curative intent in MAASTRO clinic in 2002-2003. They will be retrieved from the appointment -IT system. For all these patients will be checked whether they are alive using the MBA (municipal base administration).
Sampling Method: Non-Probability Sample
Enrollment: 387 (Actual)
Dates: Start 2013-03; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is the incidence and severity of locoregional late toxicity at 10 years after radiotherapy. | One assessment approximately 10 years after radiotherapy
  As primary endpoint, for each patients the STAT score will be determined, summarizing locoregional late toxicity, e.g. fibrosis, cosmetic outcome, shoulder dysfunction, lymphedema arm, pain [Barnett et al, 2012].

SECONDARY OUTCOMES:
The secondary endpoint is 10 year survival rate and the incidence and severity of other than locoregional late toxicity. | One assessment approximately 10 years after radiotherapy
  The secondary endpoint is 10 year survival rate, and late toxicity, other than locoregional late toxicity, e.g. fatigue, neuropathy, menopausal symptoms, cardiac and pulmonary symptoms, and secondary tumors. Survival will be divided in overall survival, locoregional recurrence free survival and distant metastases free survival. For each patient other toxicity at 10 year will be scored according to CTC-AE 4.

OTHER OUTCOMES:
In addition, we will record potential risk factors for the several outcome parameters | one consultation by physician (assistant) ten years after radiotherapy
  The following the potential risk factors are recorded:
  1. Patient related risk factors:
     * Age at time of diagnosis
     * Genetic and protein profile blood samples (optional with informed consent of participant)
     * Smoking
  2. Treatment related factors:
     * Type of surgery
     * Excision volume
     * Post-operative complications
     * Resection margins Free
     * Scar visibility
     * Axillary surgery
     * Radiotherapy
     * Fractionation scheme
     * Target volumes
     * Dose-volume parameters
     * Actually delivered dose
     * Chemotherapy
     * Hormonal treatment
     * Immunotherapy
  3. Tumor related factors
     * Localization
     * Stage
     * Differentiation grade
     * Hormonal receptors
     * HER-2
     * Genetic profile

CONTACTS AND LOCATIONS:
Overall Officials: Liesbeth J Boersma, M.D., Ph.D., Principal Investigator — Maastro Clinic, The Netherlands
Locations (1):
- MAASTRO clinic, Maastricht, Limburg, Netherlands